CLINICAL TRIAL: NCT01881204
Title: Hesperidin and Bone Health in Postmenopausal Women
Acronym: Hesperidin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Nestec Ltd. (Industry)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 10.21.NRC
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Hesperidin; Osteoporosis; Bone Loss
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic | interventions — Hesperidin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hesperidin and Calcilock (Experimental): Subjects will consume 4 cookies containing Hesperidin and Calcilock.
  Interventions: Dietary Supplement: Hesperidin and Calcilock
- Hesperidin (Experimental): Subjects will consume 4 cookies containing Hesperidin, 552mg, daily
  Interventions: Dietary Supplement: Hesperidin
- Control (Placebo Comparator): Subjects will consume 4 cookies daily without Hesperidin or Calcilock.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Hesperidin and Calcilock — Hesperidin (552mg) and Calcilock® (amount per day: Calcium: 684 mg; Phosphorus: 282mg; Magnesium: 102mg; Zinc: 2.86mg; Vitamin C: 20 mg; Vitamin K1: 28µg; Vitamin D: 1.86µg) will be administered in the form of cookies (biscuit).
  Arms: Hesperidin and Calcilock
Dietary Supplement: Hesperidin — Hesperidin (552mg) will be administered in the form of cookies (biscuit).
  Arms: Hesperidin
Dietary Supplement: Control — Cookies without Hesperidin or Calcilock added.
  Arms: Control

SUMMARY:
The primary objective of this clinical trial is to test hesperidin with and without CALCILOCK® for bone resorption suppressing effect in postmenopausal women. The secondary objective is the comparison between 41Ca technology and classical biomarker to evaluate bone resorption.

DETAILED DESCRIPTION:
Subjects will participate in four phases of the study: Baseline of 50 days and three intervention phases which include 50 days receiving product followed by 50 days of recovery. The total duration of the study will be 350 days. If participant has not been previously labeled with 41Ca, a 150 day period is added to the study.

Hesperidin (552mg) and Calcilock® (amount per day: Calcium: 684 mg; Phosphorus: 282mg; Magnesium: 102mg; Zinc: 2.86mg; Vitamin C: 20 mg; Vitamin K1: 28µg; Vitamin D: 1.86µg) will be administered in the form of cookies (biscuit).

ELIGIBILITY:
Inclusion Criteria:

* Women at least 4 years postmenopausal

Exclusion Criteria:

* Medications affecting bone resorption

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Elimination of 41Calcium in Urine. | 50 days
  Appearance of Ca41 in urine will be measured by Accelerator Mass Spectrometry to represent calcium that is being lost from the skeleton.

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, Ph.D., Principal Investigator — Purdue University; Berdine R Martin, PhD, Study Director — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Martin BR, McCabe GP, McCabe L, Jackson GS, Horcajada MN, Offord-Cavin E, Peacock M, Weaver CM. Effect of Hesperidin With and Without a Calcium (Calcilock) Supplement on Bone Health in Postmenopausal Women. J Clin Endocrinol Metab. 2016 Mar;101(3):923-7. doi: 10.1210/jc.2015-3767. Epub 2016 Jan 11. PMID 26751193